CLINICAL TRIAL: NCT01793883
Title: A Phase 2 Randomized, Double Blind, Placebo Controlled, Parallel Arm Study to Investigate the Efficacy and Safety of Inhaled Laninamivir Octanoate TwinCaps® Dry Powder Inhaler in Adults With Symptomatic Influenza A or B Infection
Brief Title: Efficacy and Safety Study of Laninamivir Octanoate TwinCaps® Dry Powder Inhaler in Adults With Influenza
Acronym: Igloo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTA51-350-201; HHSO100201100019C (Other Grant/Funding Number: HHS BARDA); 2013-000582-36 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-18 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Influenza Laninamivir Octanoate
MeSH Terms: conditions — Influenza, Human | interventions — laninamivir; CS 8958; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 40 mg Laninamivir Octanoate DPI (Active Comparator): 40 mg Laninamivir Octanoate and matching placebo
  Interventions: Drug: 40 mg Laninamivir Octanoate; Drug: Placebo
- 80 mg Laninamivir Octanoate DPI (Active Comparator): 80 mg Laninamivir
  Interventions: Drug: 80 mg Laninamivir Octanoate
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 40 mg Laninamivir Octanoate
  Other Names: CS-8958
  Arms: 40 mg Laninamivir Octanoate DPI
Drug: 80 mg Laninamivir Octanoate
  Other Names: CS-8958
  Arms: 80 mg Laninamivir Octanoate DPI
Drug: Placebo
  Other Names: Lactose
  Arms: 40 mg Laninamivir Octanoate DPI; Placebo

SUMMARY:
This Phase 2 protocol is designed to compare two dose levels of laninamivir octanoate versus placebo. The objectives are to obtain safety and efficacy in adults aged 18 to 64 years who present to clinic with symptomatic presumptive influenza A or B infection.

DETAILED DESCRIPTION:
Approximately 636 subjects will be randomized into the Study.

Following confirmation of circulating influenza in the local area, eligible subjects with recent onset of symptomatic presumptive influenza A or B infection will be enrolled in the study. Subjects must be randomized within 40 hours of the first symptom onset. Subjects will be randomized to placebo, 40 or 80 mg of laninamivir octanoate.

The study will be conducted on an outpatient basis. The first dose of study drug will be administered via inhalation within 4 hours of randomization in the clinic, followed by a second dose at home. Participants will be followed for 14 days to assess efficacy, virology and safety. Outpatient visits to the investigational site are scheduled on Days 2 (optional PK Sub-study Visit) 3, 5, 8, 15. An End of study visit will be performed on Day 29.

ELIGIBILITY:
Main Inclusion Criteria:

1. Provide written informed consent
2. Males or females aged 18-64 years, inclusive
3. Symptomatic presumptive influenza A or B infection defined as the presence of:

   1. a fever of ≥38.0ºC (≥100.4 ºF) at the screening visit OR a history of fever within the 24 hours prior to the screening visit and has administered antipyretic(s) in the 6 hours prior to the screening visit AND
   2. ≥1 moderate systemic symptom (headache, feeling feverish, body aches and pains, and fatigue) AND
   3. ≥1 moderate respiratory symptom (cough, sore throat and nasal congestion)
4. Onset of illness no more than 40 hours prior to randomization. Onset of illness is defined as the time, the first of any one of the following, occurred:

   1. time when the subjects' temperature was measured as elevated (≥38.0°C (≥100.4ºF) OR
   2. time when the subject first experienced at least one respiratory symptom (cough, sore throat and nasal congestion) OR
   3. time when the subject first experienced at least one systemic symptom (headache, feeling feverish, body aches and pains, and fatigue)

Main Exclusion Criteria:

1. Use of antiviral treatment for influenza (e.g. zanamivir, oseltamivir, rimantadine, or amantadine) within 14 days prior to screening
2. Received live attenuated or trivalent inactivated influenza virus vaccine in the previous 3 weeks.
3. History or presence of clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, cystic fibrosis, or bronchiectasis) or asthma
4. History of congestive heart failure with symptoms consistent with New York Heart Association Class III or IV functional status (See Appendix A: ) within the past 12 months
5. Presence of an immune compromised status due to chronic illness, organ transplantation or use of daily systemic immunosuppressants
6. Presence of clinically significant signs of acute respiratory distress during screening
7. Current use of inhaled medications (nasal or oral) or anticipated use of inhaled medications (nasal or oral) at any time during the study.
8. Current or a history of acute or chronic renal impairment requiring hemodialysis and/or a known or calculated creatinine clearance (CLCR) of <60 mL/min
9. History or presence of any clinical condition or evidence of organ dysfunction on examination which, in the opinion of the investigator, may affect either the subject's ability to participate in the study or the study results

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 639 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lambert, PhD, Study Director — Biota Scientific Management Pty Ltd
Locations (221):
- United States (70):
  - Scottsboro Quick Care Clinic, Scottsboro, Alabama
  - Clinical Trial Connection, Camp Verde, Arizona
  - Warner Family Practice, Chandler, Arizona
  - Clinical Research Connections, LLC, Harrisburg, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - eStudySite, Chula Vista, California
  - Beach Physicians Medical Group, Inc., Huntington Beach, California
  - eStudySite, La Mesa, California
  - Novo Research, Inc., Long Beach, California
  - Lucita M. Cruz, MD, Inc, Norwalk, California
  - eStudySite, Oceanside, California
  - Clinical Trials of Orange County, Inc, Orange, California
  - California Research Foundation, San Diego, California
  - San Diego Sports Medicine & Family Health Center, San Diego, California
  - Orange County Research Center, Inc, Tustin, California
  - SC Clinical Research, Inc., Upland, California
  - Complete Family Care, Northglenn, Colorado
  - BRCR Medical Center, Inc DBA Boca Raton Clinical Research, Boca Raton, Florida
  - Zasa Clinical Research, LLC, Boynton Beach, Florida
  - Southeast Clinical Research, LLC, Chiefland, Florida
  - Sanitas Research, Coral Gables, Florida
  - Southeast Clinical Research, LLC - Parent, Jacksonville, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - New Horizon Research Center, Inc, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - DCT - FMC, LLC, d/b/a Discovery Clinical Trials, Orlando, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Dr. B. Abraham, PC, Snellville, Georgia
  - Women's Healthcare Associates P.A., Idaho Falls, Idaho
  - Baptist Health Clinical Studies, Madisonville, Kentucky
  - Clinical Trials Management, LLC, Mandeville, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Medipharmics, LLC, Metairie, Louisiana
  - KAMP Medical Research, Natchitoches, Louisiana
  - Paul Shapero, MD, Bangor, Maine
  - Bethesda Allergy, Asthma & Research Center, LLC, Bethesda, Maryland
  - Neccr Imca, Llc, Fall River, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Oakland Medical Research Center, Troy, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - The Asthma & Allergy Center, P.C. master, Bellevue, Nebraska
  - Beacom Family Health Connection, Fremont, Nebraska
  - eStudySite, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Sentral Clinical Research Services, LLC, Cincinnati, Ohio
  - Hometown Urgent Care & Occupational Health, Milford, Ohio
  - ProMedica Health System, Inc, Sylvania, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Detweiler Family Medicine & Associates, Lansdale, Pennsylvania
  - Warminster Medical Associates, PC, Warminster, Pennsylvania
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Clinical Research Solutions, PC, Columbia, Tennessee
  - HCCA Clinical Research Solutions, Franklin, Tennessee
  - Clinical Research Solutions, PC, Franklin, Tennessee
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Clinical Research Solutions, PC, Nashville, Tennessee
  - Clinical Research Solutions, PC, Smyrna, Tennessee
  - ACRC Trials, Plano, Texas
  - Sun Research Institute, LLC, San Antonio, Texas
  - Oakwell Clinical Research, San Antonio, Texas
  - DBA Southwest Clinic, San Antonio, Texas
  - DCT-Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Westside Medical, Clinton, Utah
  - Focus Clinical Research, Draper, Utah
  - J. Lewis Research - FirstMed East, Salt Lake City, Utah
  - Carilion Infectious Disease, Roanoke, Virginia
- Australia (10):
  - Dr Doong's Surgery, Burwood, New South Wales
  - Hyde Park Medical, Sydney, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Cairns Base Hospital, Cairns, Queensland
  - Jimboomba Junction Family Practice & Skin Cancer Clinic, Jimboomba, Queensland
  - Mermaid Beach Medical Centre, Mermaid Beach, Queensland
  - Morayfield 7 Day Medical Centre, Morayfield, Queensland
  - AusTrials Pty Ltd. Sherwood, Sherwood, Queensland
  - Pain & Anaesthesia Research Clinic, Adelaide, South Australia
  - Hunter Clinical Research, Broadmeadows, Victoria
- Belgium (9):
  - Dokter Luc Timmermans, Borgerhout
  - Vereecken Guy, Halen
  - Calozet, Yven, Herbeumont
  - Hutsebaut, Andre, Moerkerke
  - Van Mulders, Norbert, Moorsel
  - Parque, Jean-Luc, Mouscron
  - Mortelmans, Jaak, Oostham
  - Private Practice, Oudenaarde
  - BVBA Dr. Luc Capiau, Wetteren
- Bulgaria (10):
  - SHATPPD-Ruse EOOD, Rousse
  - DCARC "Hill Clinic", Sofia
  - Diagnostic Consultative Center II - Sofia OOD, Sofia
  - Fifth MHAT-Sofia, EAD, Sofia
  - MHAT "Lyulin", EAD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - NMTH "Tsar Boris III", Sofia
  - UMHAT " Alexandrovska" EAD, Sofia
  - UMHAT 'Lozenets", Sofia
  - MDHAT Dr Stefan Cherkezov, AD, Veliko Tarnovo
- Canada (5):
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Etobicoke, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Omnispec Clinical Research Inc, Mirabel, Quebec
  - Clinique Medicale St-Louis (Recherche) Inc, Québec
- Colombia (3):
  - Administradora Country S.A., Bogotá
  - Centro de Investigacion Clinica - CAFAM, Bogotá
  - Clinica Colsanitas S.A. sede Clinica Universitaria Columbia, Bogotá
- Estonia (9):
  - Vee Family Doctor's Center OY, Paide
  - Medicum Perearstikeskus AS, Tallinn
  - Meie Tervis OU, Tallinn
  - Merekivi Perearstid OU, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - Mustamae Health Centre, Tallinn
  - Pirita Family Doctors Centre, Tallinn
  - Dr Monika Vask Ltd., Tartu
  - Marje Toom Family Doctors Practice, Võru
- France (8):
  - Cabinet Medical, La Bouëxière, Ille Et Vilaine
  - Cabinet Medical, Tours, Indre Et Loire
  - Cabinet Medical, La Montagne, Loire Atlantique
  - Cabinet Medical - Alain Boye, Nantes, Loire Atlantique
  - Cabinet Medical, Briollay, Maine Et Loire
  - Cabinet Medical Jacques Marty, Mûrs-Erigné, Maine Et Loire
  - Cabinet Medical Jean Charcot, Segré, Maine Et Loire
  - Cabinet Medical, Vihiers
- Germany (11):
  - Institut fuer Praeventive Medizin Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. med. Reinhold Jerwan-Keim, Renate Metz, Dietzenbach, Hesse
  - Gemeinschaftspraxis Dres. Hagemann, Duerfeld und Breiderhoff, Essen, North Rhine-Westphalia
  - Hausarztzentrum Bocholder Strasse, Essen, North Rhine-Westphalia
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - Unterfrintroper Hausarztzentrum, Essen, North Rhine-Westphalia
  - medicoKIT, Goch, North Rhine-Westphalia
  - Gemeinschaftspraxis Heisters und Sungen, Kamp-Lintfort, North Rhine-Westphalia
  - Gemeinschaftspraxis Dres. Kleinecke-Pohl, Kirsch, Benner-Hemsen, Koein, North Rhine-Westphalia
  - ABX-CRO advanced pharmaceuticals Forschungsqesellschaft mbH, Dresden, Saxony
  - Praxis Dr. Schiewe, Hamburg
- Hungary (11):
  - Clinexpert Egeszsegugyi Szolg. es Ker. Kft., Budapest
  - CSALADGYOGYYASZ Szolgaltato es Oktato Bt., Budapest
  - Haziorvosi Rendelo, Budapest
  - QUALICLINIC Eu-i Szolg. es Kutatasszervezo Kft, Budapest
  - Kenezy Korhaz es Rendelointezet, Debrecen
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Felnott Haziorvosi Rendelo, Kecskemét
  - Haziorvosi Rendelo, Kecskemét
  - Felnott Haziorvosi Rendelo, Miskolc
  - Revamed Kft., Nyíregyháza
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Latvia (8):
  - Liga Kozlovska Family Doctor Practice, Balvi
  - Jelgava Outpatient Clinic, Jelgava
  - Dr. R. Eglite's Private Practice, Kuldīga
  - Dr. Dz.Trosk's practice, Lielvārde
  - Regional Hospital of Liepaja, Liepāja
  - Hospital of Reseknes, Rēzekne
  - Clinic of GP A.Lasmanis "ALMA", Riga
  - Vecverdina Vizma - GP Practice, Riga
- Mexico (13):
  - Centro de Investigacion Medico Biologica y Terapia Avanzada (CIMBYTA), Guadalajara, Jalisco
  - Hospital de Especialidades Centro Medico Puerta de Hierro, Zapopan, Jalisco
  - Centro de Investigacion Clinica Acelerada, S.C., Mexico City, Mexico City
  - Centro de Investigacion Clinica GRAMEL S.C, Mexico City, Mexico City
  - Facultad Mexicana de Medicina, Universidad La Salle A.C., Mexico City, Mexico City
  - Hospital Angeles Lindavista, Mexico City, Mexico City
  - Mexico Centre for Clinical Research S.A. de C.V, Mexico City, Mexico City
  - Centro de Investigaction y Transferencia en Salud del Tecnologico de Monterrey, Monterrey, Nuevo León
  - Hospital Universitario de Monterrey, Monterrey, Nuevo León
  - Phylasis Clinicas Research S de RL de CV, Cuautitlán Izcalli, State of Mexico
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Nucleo Victoria de Investigacion Clinica S.C., Durango
  - Oaxaca Site Management Organization S.C., Oaxaca City
- New Zealand (5):
  - Optimal Clinical Trials, Auckland
  - Primorus Clinical Trials Ltd, Christchurch
  - Shirley Medical Centre, Christchurch
  - Clinical Trials New Zealand Ltd, Hamilton
  - Auckland Family Medical Centre, Remuera
- Peru (6):
  - Hospital Nacional Carlos Alberto Seguin Escobedo, Arequipa
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Clinica Internacional Sede San Borja, Lima
  - Clinica San Borja, Lima
  - Hospital Maria Auxiliadora, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
- South Africa (36):
  - Global Clinical Trials PE, Port Elizabeth, Eastern Cape
  - Iatros International, Bloemfontein, Free State
  - Josha Research, Bloemfontein, Free State
  - Drs YAK Vahed and Partners, Welkom, Free State
  - Maphutha, MB, Johannesburg, Gauteng
  - Medicross Roodepoort Clinical Research, Johannesburg, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - DJW Research, Krugersdorp, Gauteng
  - Synexus SA, Stanza Bopape Clinical Research Centre, Mamelodi East, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - Engelbrecht, I, Pretoria, Gauteng
  - Global Clinical Trials Pretoria, Pretoria, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Synexus SA - Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Syzygy Clinical Research Services Wilgers, Pretoria, Gauteng
  - University of Pretoria Clinical Research Unit, Pretoria, Gauteng
  - De Villiers Clinical Trials, Durban, KwaZulu-Natal
  - Sebastian, Peter, Durban, KwaZulu-Natal
  - Synapta Clinical Research, Durban, KwaZulu-Natal
  - van Rensburg, CJJ, Durban, KwaZulu-Natal
  - Vawda, ZFA, Durban, KwaZulu-Natal
  - Aliwal Shoal Medical Centre, eMkhomazi, KwaZulu-Natal
  - Brookdale Clinical Research Centre, Phoenix, KwaZulu-Natal
  - Richards Bay Trial Centre (Pty) Ltd, Richards Bay, KwaZulu-Natal
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - Mzansi Ethical Research Centre, Middelburg, Mpumalanga
  - Africa International Research, Cape Town, Western Cape
  - Allergy Diagnostic & Clinical Research Unit, Cape Town, Western Cape
  - Boyd, WV, Cape Town, Western Cape
  - Helderberg Clinical Trials Centre, Cape Town, Western Cape
  - Langeberg Clinical Trials, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Western Cape Clinical Trials, Cape Town, Western Cape
  - Excellentis Clinical Trial Consultants, George, Western Cape
  - Somerset West Clinical Trial Unit, Somerset West, Western Cape
  - Clinical Projects Research SA (PTY) LTD, Worcester, Western Cape
- United Kingdom (7):
  - Staploe Medical Centre, Ely, Cambridgeshire
  - Avondale Surgery Research, Chesterfield, Derbyshire
  - Knowle House Surgery, Plymouth, Devon
  - Sheepcot Medical Centre, Watford, Hertfordshire
  - CPS Ltd, Glasgow, Strathclyde
  - Holbrook Lane Surgery, Coventry, Warwickshire
  - Bradford on Avon Health Centre, Bradford-on-Avon, Wiltshire

RESULTS

PARTICIPANT FLOW:
Groups:
- 40 mg Laninamivir Octanoate DPI: 40 mg Laninamivir Octanoate and matching placebo
  40 mg Laninamivir Octanoate
  Placebo
- 80 mg Laninamivir Octanoate DPI: 80 mg Laninamivir
  80 mg Laninamivir Octanoate
- Placebo: Matching Placebo
  Placebo
Period: Overall Study
Arm/Group | 40 mg Laninamivir Octanoate DPI | 80 mg Laninamivir Octanoate DPI | Placebo
Started | 213 | 214 | 212
Completed | 201 | 204 | 204
Not Completed | 12 | 10 | 8
Not completed — Withdrawal by Subject | 3 | 7 | 3
Not completed — Subject noncompliance | 0 | 1 | 1
Not completed — Lost to Follow-up | 5 | 1 | 3
Not completed — Randomized in error | 1 | 0 | 0
Not completed — Unable to complete spriometry | 1 | 0 | 0
Not completed — Unable to complete measurements | 1 | 0 | 0
Not completed — Met exclusion criteria | 1 | 0 | 0
Not completed — Dosing error | 0 | 1 | 0
Not completed — Respiratory distress during spirometry | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population - all subjects who provided informed consent for this study and who had been randomized to the study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg Laninamivir Octanoate DPI | 80 mg Laninamivir Octanoate DPI | Placebo | Total
Number analyzed (Participants) | 213 | 214 | 212 | 639
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.95) | 39.2 (12.49) | 40.3 (13.31) | 39.3 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 128 | 115 | 362
  Male | 94 | 86 | 97 | 277
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 1 | 1 | 3
  United States | 102 | 97 | 84 | 283
  United Kingdom | 1 | 0 | 0 | 1
  New Zealand | 2 | 4 | 3 | 9
  Canada | 2 | 2 | 3 | 7
  Latvia | 1 | 3 | 4 | 8
  Belgium | 13 | 8 | 14 | 35
  Mexico | 7 | 12 | 10 | 29
  South Africa | 40 | 38 | 39 | 117
  Bulgaria | 27 | 32 | 36 | 95
  Germany | 6 | 4 | 3 | 13
  Estonia | 11 | 13 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of Influenza Symptoms
Description: Time to alleviation of influenza will be assessed through Flu-iiQ (Influenza intensity and impact Questionnaire) and diary cards from Day 1 to 14.
Time Frame: Efficacy will be assessed over 14 days post-randomization.
Population: Intent-to-treat-infected (ITT-I) population - all ITT subjects with laboratory confirmed influenza A or B infection by at least one virological method (qRT-PCR or qCulture) on either Day 1 or 3
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | 40 mg Laninamivir Octanoate DPI | 80 mg Laninamivir Octanoate DPI | Placebo
Number analyzed (Participants) | 67 | 75 | 89
hours | 102.30 [80.60 to 114.80] | 103.20 [89.00 to 138.30] | 104.10 [93.00 to 140.70]
Statistical Analysis 1: Comparison: 40 mg Laninamivir Octanoate DPI vs Placebo; Test type: Superiority; p = 0.251, Log Rank
Statistical Analysis 2: Comparison: 80 mg Laninamivir Octanoate DPI vs Placebo; Test type: Superiority; p = 0.818, Log Rank

ADVERSE EVENTS:
Time Frame: Period of time was defined as from Day 1 to Day 15.
Description: All-Cause Mortality data was collected for all randomized participants. Serious Adverse Events and Other (Not Including Serious) Adverse Events were collected for the Safety Analysis Set, which was defined as all patients who received at least 1 dose of study drug and had at least 1 safety assessment after randomization.
Groups:
- 80 mg Laninamivir Octanoate DPI: 80 mg Laninamivir Octanoate
  80 mg Laninamivir Octanoate
Arm/Group | 40 mg Laninamivir Octanoate DPI | 80 mg Laninamivir Octanoate DPI | Placebo
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/214 | 0/212
Serious Adverse Events (participants affected / at risk) | 1/212 | 1/211 | 1/211
Other Adverse Events (participants affected / at risk) | 31/212 | 27/211 | 21/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg Laninamivir Octanoate DPI (N=212) | 80 mg Laninamivir Octanoate DPI (N=211) | Placebo (N=211)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg Laninamivir Octanoate DPI (N=212) | 80 mg Laninamivir Octanoate DPI (N=211) | Placebo (N=211)
Bronchitis bacterial (Infections and infestations) | 6 | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 2
Headache (Nervous system disorders) | 7 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes